CLINICAL TRIAL: NCT06382714
Title: Efects of Virtual Museum Visit on Dialysis Symptoms and Anxiety in Hemodialysis Patients
Brief Title: Virtual Museum Visit on Dialysis Symptoms and Anxiety in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Mukadder Mollaoğlu, Prof.Dr, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-12/13
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-04

CONDITIONS: DIALYSIS SYMPTOMS AND ANXIETY

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy Intervention Group (Experimental): A total of five sessions of museum visits will applied to the patients in the intervention group, lasting 20-30 minutes during dialysis. The scales will administered to the individuals in the intervention groups three times in total.
  The intervention group is the group in which museum visit will applied. They receives 3 sessions of hemodialysis per week.
  Interventions: Other: For the intervention group, a museum visit with virtual reality glasses will be applied.
- Control Group (No Intervention): No virtual museum visit was applied to the control group. Scales were applied to individuals. For the control group, evaluations were made with scales three times in total.

INTERVENTIONS:
Other: For the intervention group, a museum visit with virtual reality glasses will be applied. — Patients will visit a museum while undergoing hemodialysis with virtual reality glasses for a total of five sessions for intervention group
  Arms: Art Therapy Intervention Group

SUMMARY:
The main purpose of dialysis used in the treatment of end-stage renal failure is; By relieving the patient from uremic symptoms, controlling excess fluid, electrolyte and acid base disorders, improving the well-being of the patients and also improving the quality of life of the patients. In addition to its contribution to the continuation of life, dialysis can significantly affect the biological and physiological balance and normal life order of patients. Some of these effects may be negative on patients. During this process, patients may frequently experience symptoms such as changes in fluid-electrolyte balance, increased fatigue, and weakness, as well as psychopathological conditions such as anxiety. In this context, it is extremely important to handle patients from a holistic perspective and keep their homeostatic balance under control during the hemodialysis process. In addition to pharmacological treatments, many integrative methods are used in the management of symptoms for reasons such as being low in cost, having fewer side effects than pharmacological treatments, and strengthening the immune system. Museum visit, one of these integrative treatment methods, has become an area of art therapy where help is received for various reasons such as coping with the symptoms of chronic diseases, reducing the side effects of medications, preventing mental depression, strengthening healthy behaviors, and avoiding tension and loss of control. In this context, the research was planned as a randomized controlled study investigating the effect of virtual museum tour on dialysis symptom index and anxiety in hemodialysis patients..T.R. The "https://sanalmuze.gov.tr" site belonging to the Ministry of Culture and Tourism will be shown to the patients five times and the virtual museum visit will be made by showing the patient's preferred museum five times among the 53 museums prepared by the General Directorate of Information Technologies of the Ministry of Culture and Tourism, and the Initiative Group, Control It will be compared with its group. Research data; It will be collected using the Patient Information Form, Dialysis Symptom Index and Beck Anxiety Scale (BAI). At the end of the study, the data will be evaluated in the SPSS program. The museum visit applied to the Intervention Group will also be applied to the control group after the study is completed, taking into account the ethical dimension.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been receiving hemodialysis treatment for at least one year, who are 18 years of age or older, who do not have difficulty in communicating, who are competent to answer all the questions, who do not have serious mental illness or mental problems, and who agree to participate in the research will be included in the study.

Exclusion Criteria:

Those who have just started hemodialysis treatment (< 1 year), those who have vision or hearing problems, those who have difficulty communicating, those under the age of 18, and those who do not want to participate in the study or want to leave will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dialysis Symptom Index (DSI) | It will take 5 weeks to collect data three times after randomization is done. The first measurement of dialyis symptom index will be done in the first week, the second measurement in the third week and the third measurement in the fifth week.
  It was developed by HD patients in order to determine the symptoms experienced by HD patients and the level of impact on the patient. The scale, developed from the Memorial Symptom Diagnosis Scale Short Form, consists of 30 items. Responses are obtained on a 5-point Likert scale. The total scale score is obtained by adding up the scores obtained. This value varies between "0-15 0". The value "0" indicates that there is no symptom. The increase in the total points given to the answers towards 150 points shows that the effect of the mentioned symptom is increasing. The internal consistency coefficient of the scale was determined as 0.84.
Beck Anxiety Scale (BAI) | It will take 5 weeks to collect data three times after randomization is done. The first measurement of Beck anxiety scale will be done in the first week, the second measurement in the third week and the third measurement in the fifth week.
  It measures the frequency of anxiety symptoms experienced by the individual. It is a Likert-type self-evaluation scale consisting of twenty-one items and scored between 0-3. A high total score indicates the level of anxiety experienced by the person. The validity and reliability of the scale was determined in our country.

CONTACTS AND LOCATIONS:
Locations (1):
- Mukadder, Mollaoğlu, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 31 Dec 2024

REFERENCES:
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Ulusoy M, Şahin N, Erkman H. Turkish Version of The Beck Anxiety Inventory: psychometric Properties. J Cognitive Psychotherapy: Int Quaterly. 1998; 12: 28-35.
- [Result] Weisbord SD, Fried LF, Arnold RM, Rotondi AJ, Fine MJ, Levenson DJ, Switzer GE. Development of a symptom assessment instrument for chronic hemodialysis patients: the Dialysis Symptom Index. J Pain Symptom Manage. 2004 Mar;27(3):226-40. doi: 10.1016/j.jpainsymman.2003.07.004. PMID 15010101